CLINICAL TRIAL: NCT01432925
Title: Timing of the Decision on Surgical Intervention for Buruli Ulcer Patients Treated With Rifampicin/Streptomycin
Brief Title: Timing of Surgical Intervention in Buruli Ulcer Patients Treated With Antibiotics
Acronym: Burulitime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: PNLUB, Ministère de la santé, Cotonou, République du Bénin. (Unknown); Laboratoire de Référence des Mycobactéries (Other Government)
Responsible Party: Principal Investigator, Ymkje Stienstra, MD PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BURULIVENI
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Mycobacterium Ulcerans Disease; Buruli Ulcer
Keywords: Buruli ulcer; Mycobacterium ulcerans; Streptomycin; Rifampicin; Functional limitations; surgery; Bénin
MeSH Terms: conditions — Buruli Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- evaluation surgical intervention at week 8 (Other)
  Interventions: Procedure: surgical intervention on Buruli ulcer
- evaluation surgical intervention at week 14 (Other)
  Interventions: Procedure: surgical intervention on Buruli ulcer

INTERVENTIONS:
Procedure: surgical intervention on Buruli ulcer — Can the need for surgical intervention be avoided by delay of the decision on surgical intervention, comparing the need on surgical intervention from time points of week 8 and week 14 (number of weeks after start of antibiotic treatment with streptomycin/rifampicin).

SUMMARY:
SUMMARY

Rationale: Buruli ulcer, caused by Mycobacterium ulcerans, is an ulcerative disease endemic in West Africa. It often leads to functional limitations. Treatment was by extensive surgery, until in 2005 gradually antibiotic treatment for eight weeks with rifampicin and streptomycin was added. Observation of Buruli ulcer lesions of limited size during antibiotic treatment showed that during treatment there is a paradoxical increase of the lesion, with a decrease of the lesion after week 14. Current WHO protocols advise to decide whether surgery is needed four weeks after the start of antibiotics. This might be too early in the healing process. The investigators hypothesize that delay in surgery is safe, and that it results in a reduction of the number of surgical interventions.

Objectives:

Primary Objective of this study is to compare the need for surgical treatment in standard timing of surgery at the end of eight weeks antimicrobial treatment with a policy to postpone surgical treatment until week 14.

Secondary Objectives are to study whether postponing surgery leads to less extensive surgery and a change in frequency of functional limitations;

Study design:

Patients will be randomized for surgery at week 8 after start of antibiotic treatment and week 14 after start of treatment. Reasons for treating doctors to decide to intervene with surgery will be according to current clinical practice and will be clearly defined in this protocol. Standard care of eight weeks of rifampicin and streptomycin will be given. All patients will be followed and lesional size using acetate sheet recordings will be used during follow-up.

Study population: Patients with a clinical picture of Buruli ulcer disease confirmed by diagnostic tests in the districts covered by the Buruli ulcer centers in Lalo and Allada, Benin. Patients who are pregnant, have a contraindication for general anaesthesia and children below three years old will be excluded. 130 Patients in each treatment arm will be included to detect a difference in percentage of patients needing surgery of 20 percent.

Main study parameters/endpoints: Primary outcome measure is the number of patients healed without surgery. Secondary outcome measures are the extent of surgery by measurement of lesional size, functional limitations after the end of treatment and one year after the start of treatment and the duration of admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical picture of Buruli ulcer disease in the districts covered by the Buruli ulcer centers in Lalo and Allada, Benin, will be included at start of antibiotic treatment.
* All stages of the disease will be included. Only patients with confirmed disease by direct microscopy following acid-fast staining or PCR will be included.

Exclusion Criteria:

* Patients not on the standard treatment of eight weeks of rifampicin and streptomycin for any reason, will be excluded from this study.
* Treatment with macrolide or quinolone antibiotics, or antituberculous medication, or immune-modulatory drugs including corticosteroids within the previous one month.
* Patients not compliant with the antibiotic therapy will be excluded as well. Non-compliance is defined as the use of < 70 % of the prescribed antibiotics.
* Patients with a contraindication for general anaesthesia are not able to participate.
* Pregnancy.
* Osteomyelitis.
* Lesion close to the eye, with preferred standard treatment to wait for effect antibiotic treatment on extent surgery.
* The BUFLS (Buruli ulcer functional limitation score) cannot be applied to children below three years and therefore will not participate.
* Patients reporting to refuse surgery at any point in the intended treatment, cannot be included.
* Any situation or condition which may compromise ability to comply with the trial procedures.
* Patients known to be HIV positive.
* Lack of willingness to give informed consent (and/or assent by parent/legal representative).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Healing without surgical intervention | one year
  measurement of lesions at follow up visit, if lesion closed-> healed.

CONTACTS AND LOCATIONS:
Overall Officials: D Agossadou, MD, Principal Investigator — Program national lutte contre la lèpre et l'ulcère de Buruli, ministère de la santé, Hospital Lalo; G Sopoh, MD PhD, Principal Investigator — Program national lutte contre la lèpre et l'ulcère de Buruli, Ministère de la Santé, Cotonou, Bénin, hospital Allada; Tjip S van der Werf, MD PhD, Principal Investigator — UMCG - internal medicine/infectious diseases; R OC Johnson, MD PhD, Principal Investigator — Cotonou, Bénin
Locations (2):
- Benin (2):
  - Buruli ulcer center Allada, Allada
  - Buruli ulcer center Lalo, Lalo

REFERENCES:
- [Result] Wadagni AC, Barogui YT, Johnson RC, Sopoh GE, Affolabi D, van der Werf TS, de Zeeuw J, Kleinnijenhuis J, Stienstra Y. Delayed versus standard assessment for excision surgery in patients with Buruli ulcer in Benin: a randomised controlled trial. Lancet Infect Dis. 2018 Jun;18(6):650-656. doi: 10.1016/S1473-3099(18)30160-9. Epub 2018 Apr 5. PMID 29605498
- [Derived] Barogui YT, Klis SA, Johnson RC, Phillips RO, van der Veer E, van Diemen C, van der Werf TS, Stienstra Y. Genetic Susceptibility and Predictors of Paradoxical Reactions in Buruli Ulcer. PLoS Negl Trop Dis. 2016 Apr 20;10(4):e0004594. doi: 10.1371/journal.pntd.0004594. eCollection 2016 Apr. PMID 27097163